CLINICAL TRIAL: NCT05490524
Title: SMART LIVING HOMES - WHOLE INTERVENTIONS DEMONSTRATOR FOR PEOPLE AT HEALTH AND SOCIAL RISKS
Brief Title: Smart Living Homes: GATEKEEPER System With Patients With Cancer and Dementia in Cyprus
Acronym: GATEKEEPER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cyprus University of Technology (Other)
Collaborators: Pancyprian Federation of Cancer Patients and Friends (Unknown)
Responsible Party: Principal Investigator, Angelos Kassianos, Lecturer, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CUT_DN_01
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Neoplasms; Cancer; Dementia
Keywords: cancer; digital health; dementia; eHealth; RCT
MeSH Terms: conditions — Neoplasms; Dementia

STUDY DESIGN:
Intervention Model Description: The Control group will receive standard health care with no technical support, where the intervention groups will receive platform and device services provided to each user. In that respect, Intervention Group 1 will receive no real-time feedback, where Intervention Group 2 will unhand with real data and notifications.
  group)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients, research assistants, nurses, social workers, physiotherapists and psychologists responsible for data collection will not have access to the information of which group (control or intervention) the participant is.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): The Control group will receive standard health care with no technical support, where the intervention groups will receive platform and device services provided to each user. In that respect, Intervention Group 1 will receive no real-time feedback, where Intervention Group 2 will unhand with real data and notifications.
  A control group is defined as a group of clinical trial participants who will not be provided any digital devices as part of the trial and will receive care as usual by PASYKAF and AMEN.
- Intervention group 1 (limited technology) (Experimental): Intervention Group 1 - platform/devices (no real feedback provided (limited technology group) A limited technology group is defined as a group of clinical trial participants who receive the digital devices but not the automated interventions through the devices (prompts, messages).
  Interventions: Device: GATEKEEPER
- Intervention group 2 (full technology) (Experimental): Intervention Group 2 -platform/devices (with real feedback provided) (full technology group) A full technology group is defined as a group of clinical trial participants who receive the digital devices as part of the trial and healthcare professionals receive the patients' data.
  Interventions: Device: GATEKEEPER

INTERVENTIONS:
Device: GATEKEEPER — The GATEKEEPER is a digital platform that allows patients and caregivers to record their day-to-day symptoms and other parameters such as quality of life using means such as apps and wearable devices that record both self-report (quality of life, depression, anxiety) and physiological data (mobility, pain, sleep patterns, heart rate), and allows healthcare professionals to monitor these data and tailor healthcare so to prevent and intervene in symptoms that may be occurring.
  Arms: Intervention group 1 (limited technology); Intervention group 2 (full technology)

SUMMARY:
The main objective of the Project is to create a GATEKEEPER, that connects healthcare providers, businesses, entrepreneurs, elderly citizens and the communities they live in, in order to originate an open, trust-based arena for matching ideas, technologies, user needs and processes, aimed at ensuring healthier independent lives for the ageing populations. By 2022, GATEKEEPER will be embodied in an open source, European, standard-based, interoperable and secure framework available to all developers, for creating combined digital solutions for personalised early detection and interventions that (i) harness the next generation of healthcare and wellness innovations; (ii) cover the whole care continuum for elderly citizens, including primary, secondary and tertiary prevention, chronic diseases and co-morbidities; (iii) straightforwardly fit "by design" with European regulations, on data protection, consumer protection and patient protection (iv) are subjected to trustable certification processes; (iv) support value generation through the deployment of advanced business models based on the VBHC paradigm.

GATEKEEPER will demonstrate its value by scaling up, during a 42-month work plan, towards the deployment of solutions that will involve ca 40.000 elderly citizens, supply and demand side (authorities, institutions, companies, associations, academies) in 8 regional communities, from 7 EU member states. Recently 3 Asian pilots have been added as a result of the Open Calls.

The achievement of the overall objective is supported by the following, among others, specific objective: To execute a series of PILOTS to demonstrate the effect, benefit, value and scalability of the GATEKEEPER solutions around REFERENCE USE CASES COVERING PRIMARY, SECONDARY and TERTIARY PREVENTION, initially deployed in 8 regions of 7 European countries.

The Cyprus pilot mainly focuses on the early detection of the condition worsening of cancer and dementia patients by monitoring whether the use of technology can trigger appropriate management, thereby reducing the need for higher acuity care, and even, at times, improving survival by supporting demand-driven solutions through high-quality health mobile systems.

DETAILED DESCRIPTION:
Primary Outcome The Primary Objective of the proposed pilot will be the improved Health-Related Quality of Life (HRQoL) for patients participating in the full intervention and limited intervention groups compared to patients in the control group.

It is hypothesized that the improvement will he higher for the full intervention group patients compared to the limited intervention group patients.

Secondary Objectives

The secondary outcomes are measured as follows:

1. Secondary Objective for patients: includes improved parameters of patients participating in the full and limited intervention groups associated with the improvement in disease self-management; symptom burden; motivation; mobility; sleep hygiene; depression and anxiety.
2. Secondary Objective for caregivers: includes improved parameters of caregivers participating in the full and limited intervention groups associated with caregiver burden; depression and anxiety.
3. Secondary Objective for healthcare professionals: includes improved parameters of healthcare professionals before and after introducing technology associated with anxiety and technology acceptance.
4. Secondary Objective for technology evaluation: includes the feasibility, usability and acceptability of the technology used by patients, caregivers and healthcare professionals.

Materials

Hardware

* Activity Tracker - Garmin Venu Sq. 37mm is a wearable watch suitable for Health Monitoring (i.e. wrist-based heart rate, daily resting heart rate, abnormal heart rate alerts, all-day stress, relaxation reminders, relaxation breathing timer, sleep)
* Tablet - LENOVO Tab M10 10.1'' 64GB
* Tablet - LENOVO Tab M10 4G LTE 10.1'' 32GB
* Mobile XIAOMI Redmi 9C

Questionnaires

There will be three evaluation periods (baseline, intermediate and final) during the two-year pilot and the evaluation tools used are the following:

Self-report at home (PASYKAF) or at inpatient and outpatient clinic (AMEN) through GATEKEEPER using tablets

Patients:

For PASYKAF

* Socio-demographics information including age, gender, educational level, marital status, type of diagnosis etc.
* EORTC QLQ C-30 (1) is a cancer health-related quality-of-life questionnaire that has been widely validated and used in clinical trials and investigations using PROs for individual patient management. It is composed of both multi-item scales and single-item measures. The QLQ-C30 will be administered at admission and at 6 weeks.
* IPOS (2) is a measure of global symptom burden which includes items that measure physical, psychosocial, social and spiritual domains in line with an impeccable holistic assessment. It allows patients to list their main concerns, to add other symptoms they are experiencing, and to state whether they have unmet information or practical needs. It can assess and monitor symptoms and concerns in advanced illness, determine the impact of healthcare interventions, and demonstrate quality of care. The IPOS will be administered at admission and at 6 weeks.
* HADS (3) is a self-report scale developed to assess psychological distress in non-psychiatric patients in both hospital and community settings. It consists of two subscales, measuring symptoms of depression (HADS-D), and anxiety (HADS-A). Following completion of the HADS, a pop-up section will follow that allows use cases to provide any additional information that they may feel is important regarding their psychological well-being - qualitative data/ free word to describe their personal lived experience (completion is optional). HADS will be administered at admission and at 6 weeks.
* System Usability Scale (SUS) (4) (simplified version) will assess the usability of the platform and the devices on a 5-point Likert scale (1 = strongly disagree and 5 = strongly agree). SUS will be administered at 6 weeks.
* The Single Ease Question (SEQ) will assess the level of difficulty for each interaction on a 7-point Likert scale (1 = very difficult and 7 = very easy). SEQ will be administered at 6 weeks.

For AMEN

* EQ-5D (5) is a standardised measure of health status to provide a simple, generic measure of health for clinical and economical appraisal. The EQ-5D provides a simple descriptive profile and a single summary index value for health status. The EQ-5D will be administered at admission and at 6 weeks.
* MOCA (Montreal Cognitive Assessment Greek Version) assess the cognitive decline of the person based on tasks related to attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The MOCA will be administered at admission and at 6 weeks.
* Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. The MMSE will be administered at admission and at 6 weeks.
* Geriatric Depression Scale (GDS) (6) will be used to measure depression and is often used to assess depression in the elderly patients. The app will utilize simple, easy to respond, and user-friendly statements or questions that can be answered by the patient or/and the main caregiver.
* Geriatric Anxiety Scale (GAS) (7) will be used to measure anxiety and is often used to assess depression in the elderly patients. The app will utilize simple, easy to respond, and user-friendly statements or questions that can be answered by the patient or/and the main caregiver.
* System Usability Scale (SUS). A simplified version of the SUS will assess the usability of the platform and the devices on a 5-point Likert scale (1 = strongly disagree and 5 = strongly agree). SUS will be administered at 6 weeks.
* The Single Ease Question (SEQ). SEQ will assess the level of difficulty for each interaction on a 7-point Likert scale (1 = very difficult and 7 = very easy). SEQ will be administered at 6 weeks.

Caregivers:

For AMEN and PASYKAF

* Zarit Burden Interview (8) is a self-report questionnaire assesses caregiver perceptions of burden that may inadvertently affect their health, personal, social or financial wellbeing.
* System Usability Scale (SUS) will assess the usability of the platform and the devices on a 5-point Likert scale (1 = strongly disagree and 5 = strongly agree).
* The Single Ease Question (SEQ) will assess the level of difficulty for each interaction on a 7-point Likert scale (1 = very difficult and 7 = very easy).
* Beck Depression Inventory (BDI) (9) is a standardized measure to assess symptoms of depression in the general population.
* State Trait Anxiety Inventory (STAI) (10) is a standardized measure to assess anxiety in the general population.

Healthcare Professionals:

For AMEN and PASYKAF

* A modified version of the Unified Theory of Acceptance and Use of Technology (UTAUT) (11,12) tool will be used to assess whether healthcare professionals accept the use of GATEKEEPER and other technologies during the study.
* System Usability Scale (SUS) will assess the usability of the platform and the devices on a 5-point Likert scale (1 = strongly disagree and 5 = strongly agree).
* The Single Ease Question (SEQ) will assess the level of difficulty for each interaction on a 7-point Likert scale (1 = very difficult and 7 = very easy).

Research Design This is a pilot randomized controlled trial (RCT) with between and within subject design

Randomization Stratified random sampling creating subgroups based on gender, age range, and stage of illness (for both organizations). We will use the ECOG scale (13) to assess cancer patients' stage. We will use a randomization at the patient 1:1 level. Nurse assistants, social workers, physiotherapists and psychologists cannot be employed in both sites at a time and patients are unlikely to move from a control to an intervention facility, due to the geographical spread of facilities and the fact that they treat different conditions (cancer at PASYKAF and dementia at AMEN). We will also audit the recruitment rates across arms to investigate the extent of any differential recruitment and if any bias might accrue. The sites will be visited by the Field Coordinator and other research staff to present the project and its needs; a consultant statistician will then produce the random allocation of patients for either the intervention or the control arm of the study.

Blinding procedures The Research Assistants, nurses, social workers, physiotherapists and psychologists responsible for data collection will not have access to the information of which group (control or intervention) the participant is.

Study Population The users involved in the pilot are cancer patients (+50) and dementia patients (+65) that face comorbidities, professional caregivers or relatives that have the role of the informal caregivers and health care professionals of the participating organizations.

In more detail:

i. Patients with mild, moderate, and severe dementia aged 60+ and high complexity level cancer patients, aged 50+, will participate in the study. People with dementia will be recruited by the "Archangelos Michael" nursing home (AMEN) and people with cancer will be recruited by the Cyprus Association of Cancer Patients and Friends (PASYKAF).

ii. Healthcare professionals from both organisations will participate in the study. This includes professions of psychologists, social workers, speech therapists, nursing staff, physiotherapists, gymnasts and art therapists (e.g., music therapists, paint therapist, theatre therapist).

iii. Two hundred and fifty cancer patients' caregivers (n=250) and one hundred and forty-five dementia patients' caregivers (n= 145) will also participate in the study.

Procedure

The intervention will be delivered at a community level as following:

The patients of both organisations will be screened to fulfil the inclusion criteria (i.e., face difficulties with co-morbidities). Then, participants (also including informal caregivers) in the intervention group will be provided with a health-promotion application based on software and hardware (commercial devices) solutions for supporting and managing users.

The Control Group will receive current standard of care for any of their ongoing health conditions. In addition to this, and following randomization, their symptomatology and quality of life will also be assessed, at least three times (in the participant's baseline assessment, and follow-ups). In each of these encounters, there are established procedures to implement appropriate action if further mental health support is needed.

Sample Size Calculation

This is a pilot RCT (14) so according to standard procedures a formal power calculation is not required and sample was determined by the research team based on experience. However, we have performed sample power calculation for patients participating in the trial as followed:

We estimated that with 251 patients, the study would have 80% power to detect a significant between-group difference in the change in the HRQOL score from baseline to 6 weeks, with a medium effect size of 0.5 SD. We allowed for the enrollment of an additional 20% of participants in order to compensate for the loss of any patients to follow-up which provides a targeted sample size of 300 patients.

Assignment to study groups The Control group will receive standard health care with no technical support, where the intervention groups will receive platform and device services provided to each user. In that respect, Intervention Group 1 will receive no real-time feedback, where Intervention Group 2 will unhand with real data and notifications.

Control Group - standard healthcare (no technology group) A control group is defined as a group of clinical trial participants who will not be provided any digital devices as part of the trial and will receive care as usual by PASYKAF and AMEN.

Intervention Group 1 - platform/devices (no real feedback provided (limited technology group) A limited technology group is defined as a group of clinical trial participants who receive the digital devices but not the automated interventions through the devices (prompts, messages).

Intervention Group 2 -platform/devices (with real feedback provided) (full technology group) A full technology group is defined as a group of clinical trial participants who receive the digital devices as part of the trial and healthcare professionals receive the patients' data.

Asessment Timeline Screening (e.g., ECOG etc.) for eligibility Baseline assessment (all questionnaires will be completed and patients and caregivers in intervention groups will receive the devices).

During the intervention (6 weeks) (self-report and physiological parameters assessment using the wearable devices and the app Follow up at 6 weeks (all questionnaires will be completed and in addition patients, caregivers and healthcare professionals in intervention groups will complete questionnaires related to usability, feasibility and acceptability of technology).

ELIGIBILITY:
Inclusion criteria (cancer patients):

* Aged: Over the age of 50 years
* Adequate understanding of Greek and/or English Language
* Cancer diagnosis/ ICD-10: Illness classification system
* Functional status/ ECOG Performance Status 0,1,2,3
* ECOG Performance Status 4 only if Phase of Illness and Prognosis permits
* Phase of illness (Based on Medical Assessment and presenting prognosis/ the Patient is expected by the Health Care Team to be able to complete the 6-week study period)
* Patient receiving Health Care Services from PASYKAF

Exclusion criteria (cancer patients):

* Aged < 50 years
* Psychiatric diagnosis

Inclusion criteria (cancer patients' caregivers):

* Over the age of 18 years
* Adequate understanding of Greek and/or English Language
* Primary caregiver of patient with cancer
* Patient/ Caregiver receiving Health Care Services from PASYKAF (The primary caregiver is a family member or friend that supports a patient through cancer treatment, helps with daily activities, such as going to the doctor or preparing meals, coordinates services and care and provides emotional and spiritual support, www.cancer.gov)

Exclusion criteria (cancer patients caregivers):

* Aged < 18 years
* Not able to consent

Inclusion criteria (healthcare professionals)

* PASYKAF employed Health Care Professionals( Nurses, Psychologists, Social Workers and Physiotherapists) that provide services in all districts of Cyprus (Nicosia, Limassol, Larnaca, Paralimni, Pafos)
* Adequate understanding of Greek and/or English Language

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Health Related Quality of Life (cancer patients only) | Baseline and follow up at 6 weeks
  EORTC QLQ C-30 is a cancer health-related quality-of-life questionnaire that has been widely validated and used in clinical trials and investigations using PROs for individual patient management. It is composed of both multi-item scales and single-item measures. The QLQ-C30 will be administered at admission and at 6 weeks. It is hypothesized that the improvement will he higher for the full intervention group patients compared to the limited intervention group patients.
Health status (dementia patients only) | Baseline and follow up at 6 weeks
  EQ-5D is a standardised measure of health status to provide a simple, generic measure of health for clinical and economical appraisal. The EQ-5D provides a simple descriptive profile and a single summary index value for health status. The EQ-5D will be administered at admission and at 6 weeks.

SECONDARY OUTCOMES:
Symptom burden (cancer patients only) | Baseline and follow up at 6 weeks
  IPOS is a measure of global symptom burden which includes items that measure physical, psychosocial, social and spiritual domains in line with an impeccable holistic assessment. It allows patients to list their main concerns, to add other symptoms they are experiencing, and to state whether they have unmet information or practical needs. It can assess and monitor symptoms and concerns in advanced illness, determine the impact of healthcare interventions, and demonstrate quality of care. The IPOS will be administered at admission and at 6 weeks.
Anxiety (cancer patients only) | Baseline and follow up at 6 weeks
  HADS is a self-report scale developed to assess psychological distress in non-psychiatric patients in both hospital and community settings. It consists of two subscales, measuring symptoms of depression (HADS-D), and anxiety (HADS-A). Following completion of the HADS, a pop-up section will follow that allows use cases to provide any additional information that they may feel is important regarding their psychological well-being - qualitative data/ free word to describe their personal lived experience (completion is optional). HADS will be administered at admission and at 6 weeks.
Depression (cancer patients only) | Baseline and follow up at 6 weeks
  HADS is a self-report scale developed to assess psychological distress in non-psychiatric patients in both hospital and community settings. It consists of two subscales, measuring symptoms of depression (HADS-D), and anxiety (HADS-A). Following completion of the HADS, a pop-up section will follow that allows use cases to provide any additional information that they may feel is important regarding their psychological well-being - qualitative data/ free word to describe their personal lived experience (completion is optional). HADS will be administered at admission and at 6 weeks.
System Usability | Follow up at 6 weeks
  System Usability Scale (SUS) (simplified version) will assess the usability of the platform and the devices on a 5-point Likert scale (1 = strongly disagree and 5 = strongly agree). SUS will be administered at 6 weeks.
System Feasibility | Follow up at 6 weeks
  The Single Ease Question will assess the level of difficulty for each interaction on a 7-point Likert scale (1 = very difficult and 7 = very easy). SEQ will be administered at 6 weeks.
Cognitive decline (dementia patients only) | Baseline and follow up at 6 weeks
  MOCA (Montreal Cognitive Assessment Greek Version) assess the cognitive decline of the person based on tasks related to attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The MOCA will be administered at admission and at 6 weeks.
Cognitive function (dementia patients only) | Baseline and follow up at 6 weeks
  Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. The MMSE will be administered at admission and at 6 weeks.
Depression (dementia patients only) | Baseline and follow up at 6 weeks
  Geriatric Depression Scale (GDS) will be used to measure depression and is often used to assess depression in the elderly patients. The app will utilize simple, easy to respond, and user-friendly statements or questions that can be answered by the patient or/and the main caregiver.
Anxiety (dementia patients only) | Baseline and follow up at 6 weeks
  Geriatric Anxiety Scale (GAS) will be used to measure anxiety and is often used to assess depression in the elderly patients. The app will utilize simple, easy to respond, and user-friendly statements or questions that can be answered by the patient or/and the main caregiver.
Caregiver burden (caregivers only) | Baseline and follow up at 6 weeks
  Zarit Burden Interview is a self-report questionnaire assesses caregiver perceptions of burden that may inadvertently affect their health, personal, social or financial wellbeing.
Depression (caregivers only) | Baseline and follow up at 6 weeks
  Beck Depression Inventory (BDI) is a standardized measure to assess symptoms of depression in the general population.
Anxiety (caregivers only) | Baseline and follow up at 6 weeks
  State Trait Anxiety Inventory (STAI) is a standardized measure to assess anxiety in the general population.
Technology acceptance (healthcare professionals only) | Baseline and follow up at 6 weeks
  A modified version of the Unified Theory of Acceptance and Use of Technology (UTAUT) tool will be used to assess whether healthcare professionals accept the use of GATEKEEPER and other technologies during the study.

OTHER OUTCOMES:
Activity tracker | Daily data for 6 weeks
  Activity Tracker - Garmin Venu Sq. 37mm is a wearable watch suitable for Health Monitoring (i.e. wrist-based heart rate, daily resting heart rate, abnormal heart rate alerts, all-day stress, relaxation reminders, relaxation breathing timer, sleep)

CONTACTS AND LOCATIONS:
Overall Officials: Angelos P. Kassianos, PhD, Principal Investigator — Cyprus University of Technology
Locations (1):
- Cyprus University of Technology, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided
The Data Sharing Agreement is underway